CLINICAL TRIAL: NCT05686044
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Multicenter Study of Buntanetap in Participants With Mild to Moderate Alzheimer's Disease
Brief Title: A Dose-ranging Study to Investigate Efficacy of Buntanetap in Mild to Moderate AD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Annovis Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANVS -22002
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer
MeSH Terms: conditions — Alzheimer Disease | interventions — phenserine

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 7.5mg Buntanetap/Posiphen (Experimental): Buntanetap/Posiphen 7.5mg oral capsule with daily administration for a period of 12 weeks
  Interventions: Drug: Buntanetap/Posiphen
- 15mg Buntanetap/Posiphen (Experimental): Buntanetap/Posiphen 15mg oral capsule with daily administration for a period of 12 weeks
  Interventions: Drug: Buntanetap/Posiphen
- 30mg Buntanetap/Posiphen (Experimental): Buntanetap/Posiphen 30mg oral capsule with daily administration for a period of 12 weeks
  Interventions: Drug: Buntanetap/Posiphen
- Placebo (Placebo Comparator): Placebo oral capsule with daily administration for a period of 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buntanetap/Posiphen — HPMC (vegetarian source) capsule shells
  Other Names: Posiphen Tartrate
  Arms: 15mg Buntanetap/Posiphen; 30mg Buntanetap/Posiphen; 7.5mg Buntanetap/Posiphen
Drug: Placebo — HPMC (vegetarian source) capsule shells
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure efficacy and safety of three different doses of buntanetap/Posiphen compared with placebo in participants with mild to moderate Alzheimer's disease.

Study details include:

The double-blind treatment duration will include a screening period of up to 42 days followed by 12 weeks of treatment at home.

The study duration will be 4-5 months. There will be 4 in-clinic visits and 1 phone call.

DETAILED DESCRIPTION:
320 mild to moderate AD participants will be randomized to 7.5 mg, 15 mg, 30mg of buntanetap/Posiphen once daily (QD) or placebo. If they provide informed consent, they will undergo a Screening Visit, and if they are considered eligible per the inclusion and exclusion criteria, they will proceed to participate in the treatment period. Randomized participants will visit the clinic for the first-time dosing in clinic, followed by an at home dosing period of 12 weeks, with daily administration of 7.5 mg, 15 mg or 30 mg of buntanetap/Posiphen or placebo. Participants will be required to visit clinics Day 0 (baseline), 6 weeks, and 12 weeks (end-of-trial), where they will undergo study procedures that include safety assessments (AE and concomitant medication monitoring, 12-lead ECGs, clinical laboratory testing, vital signs assessments, and physical examinations) and psychometric tests (Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog11), Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC), Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living Scale (ADCS-ADL), Digital Symbol Substitution Test (DSST), Mini Mental State Examination (MMSE)). At the end of blood sampling, the participants will need to stay for a minimum of 1 hour of observation. After all end-of-study procedures are complete, the subject will be discharged to home. A 24-hour follow-up call will occur after all clinical visits to assess the participants current condition and if there are any additional adverse events or questions.

The study will be a 12-weeks, placebo-controlled and double-blind trial: participants, investigators and the sponsor will be blinded to the participants' treatment.

Qualified participants will be randomly assigned at a 1:1:1:1 ratio to one of the four treatment arms: buntanetap/Posiphen 7.5 mg, buntanetap/Posiphen 15 mg, buntanetap/Posiphen 30mg, and placebo, through an Interactive Randomization System, after a screening period of up to 42 days.

ADAS-Cog 11, ADCS-CGIC, ADCS-ADL, DSST, and MMSE will be assessed by clinicians who have successfully completed the requisite certifications/trainings for each assessment.

One interim analysis is planned. It will take place when 90 enrolled subjects (~30%) have completed the Week 6 assessments to re-assess the sample size. No interim analyses are planned for the purpose of stopping the study early for futility.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Alzheimer's disease according to National Institute on Aging and National Institute on Aging and Alzheimer's Association criteria for probable AD
2. Male or female aged 55 - 85 years.
3. MMSE 14-24.
4. Have a study partner who will provide written informed consent to participate, is in frequent contact with the participant (defined as at least 10 hours per week) and will accompany the participant to study visits at designated times.
5. Female participants of childbearing potential* must have a negative urine pregnancy test at Screening, must be non-lactating and must agree to use a highly effective method of contraception (i.e., a method resulting in a failure rate of less than 1% per year when used consistently and correctly) during the trial and for 4 weeks after the last dose of trial treatment, such as:

   * Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation
   * Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Vasectomized partner (a vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the participant, and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used)
   * Sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be in relation to the duration of the study and the preferred and usual lifestyle of the participant) *Non-childbearing potential includes surgically sterilized or postmenopausal with no menstrual bleeding for at least one year prior to study start.
6. Male participants must be sterile or sexually inactive or agree not to father a child during the study and one month after the last dose of study medication and must agree to use a barrier method for contraception. Female partners of male subject must adopt a highly effective method of contraception with a failure rate of less than 1% per year when used consistently and correctly such as:

   * Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation
   * Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
7. Participants can provide written informed consent. If PI deems that participant cannot fully understand the consent form to give consent, their legally authorized representative (LARs) can provide written informed consent. Participants can comply with scheduled visits, and other study-related procedures to complete the study with the help of the study partner.
8. No evidence of current suicidal ideation or previous suicide attempt in the past 2 months as evaluated in the Columbia Suicide Severity Rating Scale nor suicidal behavior in the past 6 months as per investigator.
9. Stability of permitted medications for at least 4 weeks prior to screening.

   1. Cholinesterase inhibitors and/or memantine medication
   2. Anticonvulsant medications used for epilepsy or mood stabilization, neuropathic pain indications.
   3. Mood-stabilizing psychotropic agents, including, but not limited to, lithium.
10. Adequate visual and hearing ability (physical ability to perform all the study assessments) as per investigator.
11. Good general health with no disease expected to interfere with the study as per investigator.

Exclusion Criteria:

1. Has a history of a psychiatric disorder such as schizophrenia, bipolar disorder or major depression according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM). Mild depression or history of depression that is stable on treatment with a selective serotonin reuptake inhibitor (SSRI) or selective norepinephrine reuptake inhibitor (SNRI) medication at a stable dose is acceptable.
2. Has non-AD dementia, such as vascular dementia, Lewy body dementia, frontotemporal disease, Parkinson disease dementia, B12 and thyroid deficiency caused dementia.
3. History of a seizure disorder, if stable on medication is acceptable.
4. Has a history or current evidence of long QT syndrome, Fridericia's formula corrected QT (QTcF) interval ≥ 450 ms for men and 460 ms for women, or torsades de pointes.
5. Has bradycardia (<50 bpm) or tachycardia (>100 bpm) on the ECG at screening.
6. Has uncontrolled Type-1 or Type-2 diabetes. A subject with HbA1c levels up to 7.5% can be enrolled if the investigator believes the subject's diabetes is under control.
7. Has clinically significant renal (CKD-EPI with normal <60 mL/min/BSA (body surface area) or hepatic impairment (ALP > 2.0 ULN and/or total bilirubin > 2.0 ULN) .
8. Has any clinically significant abnormal laboratory values. Participants with liver function tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than twice the upper limit of normal will be excluded.
9. Is at imminent risk of self-harm, based on clinical interview and responses on the C SSRS, or of harm to others in the opinion of the Investigators. Participants must be excluded if they report suicidal ideation with intent, with or without a plan or method (e. g. positive response to Items 4 or 5 in assessment of suicidal ideation on the C SSRS) in the past 2 months, or suicidal behavior in the past 6 months.
10. Has cancer or has had a malignant tumor within the past year, except participants who underwent potentially curative therapy with no evidence of recurrence. (Participants with stable untreated prostate cancer or skin cancers are not excluded).
11. Alcohol / Substance use disorder, moderate to severe, in the last 5 years according to the most current version DSM.
12. Participation in another clinical trial with an investigational agent and have taken at least one dose of study medication, unless unblinded on placebo, within 4 weeks prior to the start of screening, or five half-lives of the investigational drug, whichever is greater.

    The end of a previous investigational trial is the date the last dose of an investigational agent was taken.
13. Participants with learning disability or developmental delay.
14. Participants whom the site PI deems to be otherwise ineligible.
15. Participants with a known allergy to the investigational drug or any of its components. Here are all the inactive ingredients of the investigational medicinal product:

    * Silicified Microcrystalline Cellulose
    * Dibasic Calcium Phosphate Dihydrate
    * Mannitol
    * Magnesium Stearate
    * Hypromellose (capsule shells structure)
    * titanium dioxide (opacifier of the capsule shells)
16. Subject is currently pregnant, breast-feeding and/or lactating.
17. Subject is currently taking strong and moderate CYP3A4 inhibitors and/or inducers. (e.g., CYP3A4 inhibitors Itraconazole, Ketoconazole, Azamulin, Troleandomycin, Verapamil; CYP3A4 inducers Rifampicin)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - CCT Research - Gilbert Neurology Partners, Gilbert, Arizona
  - CCT Research - Foothills Center, Phoenix, Arizona
  - The Belinga Clinic, Fort Smith, Arkansas
  - Sun Valley Research Center, Imperial, California
  - CenExel Clinical Clinical Research, Inc, Los Alamitos, California
  - Cenexel Rocky Mountain Clinical Research, Englewood, Colorado
  - Ki Health Partners LLC D/B/A New England Institute for Clinical Research, Stamford, Connecticut
  - Visionary Investigators Network, Aventura, Florida
  - K2 Medical Research, Clermont, Florida
  - The Neurology Institute - Coral Springs, Coral Springs, Florida
  - JY Research Inst., Cutler Bay, Florida
  - Arrow Clinical trial, Daytona Beach, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - New Life Medical Research Center, Hialeah, Florida
  - CenExel RCA, Hollywood, Florida
  - Coral Clinic Reserach LLC, Homestead, Florida
  - Charter Research, Lady Lake, Florida
  - ClinCloud, LLC, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - Merritt Island Clinical Research LLC, Merritt Island, Florida
  - Premier Clinical Research Institute, Inc, Miami, Florida
  - Gold Coast Health Research, LLC, Miami, Florida
  - Medical Professional Clinical Research Center, Inc, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Ezy Medical Research Co., Miami, Florida
  - Nuovida Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Visionary Investigators Network, Pembroke Pines, Florida
  - Napa Research, Pompano Beach, Florida
  - K2 Medical Research, Tampa, Florida
  - K2 Summit Research, The Villages, Florida
  - ClinCloud, LLC, Viera, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Charter Research, Winter Park, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Hawaii Pacific Neuroscience, LLC, Honolulu, Hawaii
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Josephson Wallack Munshower Neurology, P.C., Indianapolis, Indiana
  - Northern Light Acadia Hospital, Bangor, Maine
  - MedVadis Research, Waltham, Massachusetts
  - Quest Research Institue, Farmington Hills, Michigan
  - Insight Research Institute, Flint, Michigan
  - Hassman Research Institute, Berlin, New Jersey
  - CenExel Clinical Research, Inc, Toms River, New Jersey
  - Velocity Clinical Research, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University, Durham, North Carolina
  - Neuroscience Centre (CINAC), Canton, Ohio
  - Dayton Center for Neurological Disorders, Inc, Centerville, Ohio
  - NeuroCare Plus, Houston, Texas
  - Be Well Clinical Studies, LLC, Round Rock, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Inland Northwest Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 7.5mg Buntanetap/Posiphen | 15mg Buntanetap/Posiphen | 30mg Buntanetap/Posiphen
Started | 89 | 88 | 87 | 87
Completed | 82 | 84 | 80 | 79
Not Completed | 7 | 4 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 7.5mg Buntanetap/Posiphen | 15mg Buntanetap/Posiphen | 30mg Buntanetap/Posiphen | Total
Number analyzed (Participants) | 89 | 88 | 87 | 87 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (6.97) | 73.6 (7.28) | 74.7 (6.06) | 73.1 (6.15) | 73.6 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 44 | 57 | 210
  Male | 37 | 31 | 43 | 30 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 33 | 32 | 43 | 144
  Not Hispanic or Latino | 53 | 55 | 55 | 44 | 207
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 7 | 6 | 5 | 7 | 25
  White | 80 | 78 | 77 | 77 | 312
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 3
Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Mini-Mental State Examination (MMSE) is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30 with a lower score indicating greater disease severity.
  units on a scale | 20.2 (3.04) | 19.6 (3.23) | 20.0 (3.06) | 20.0 (2.82) | 20.0 (3.04)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in ADAS-Cog11
Description: Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog11) measures cognitive functions and non-cognitive functions such as mood and behavior. It was designed to measure the cognitive and behavioral domains known to be affected in Alzheimer disease, including memory, language, orientation, construction, and planning of simple designs, and completed simple goal-oriented behaviors.
  Specifically, the ADAS-Cog comprises ratings from 11 components: word recall, word recognition, constructional praxis, orientation, naming objects and fingers, commands, ideational praxis, remembering test instructions, spoken language, word finding, and comprehension.
  Total scores range from 0-70, with higher scores indicating greater cognitive impairment.
Time Frame: Baseline to the end of treatment period (12 weeks)
Population: Participants with ADAS-Cog11 scores at Baseline and 12 weeks (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 7.5mg Buntanetap/Posiphen | 15mg Buntanetap/Posiphen | 30mg Buntanetap/Posiphen
Number analyzed (Participants) | 79 | 81 | 78 | 79
units on a scale | -2.32 (0.533) | -1.34 (0.526) | -3.01 (0.534) | -2.24 (0.531)

2. Primary Outcome: ADCS-CGIC at Week 12
Description: Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) focuses on clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the patient and interview of informants.
  The ADCS-CGIC measures whether the effects of active treatment are substantial enough to be detected by a skilled and experienced clinician on the basis of a clinical interview and examination. It relies on both direct examination of the patient and an interview of the study partner.
  A skilled and experienced clinician who is blinded to treatment assignment rates the patient on a 7-point Likert scale, ranging from 1 (marked improvement) to 7 (marked worsening). Lower scores indicate better improvement.
Time Frame: Baseline to the end of treatment period (12 weeks)
Population: Participants with ADCS-CGIC scores at Baseline and 12 weeks (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 7.5mg Buntanetap/Posiphen | 15mg Buntanetap/Posiphen | 30mg Buntanetap/Posiphen
Number analyzed (Participants) | 82 | 84 | 80 | 79
score on a scale | 3.58 (0.129) | 3.96 (0.128) | 3.61 (0.131) | 3.83 (0.132)

3. Secondary Outcome: Change From Baseline to Week 12 in ADCS-ADL
Description: Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living Scale (ADCS-ADL) is a 23-item inventory scale developed as a rater-administered questionnaire answered by the participant's study partner.
  The ADCS-ADL measures 6 basic activities of daily living (BADL) items and 17 instrumental activities of daily living (IADL) items that provide a total score from 0-78, with a lower score indicating greater severity. Basic activities include basic self-care tasks such as feeding, mobility, toileting, bathing, grooming and dressing. Instrumental activities are more complex and vary based on cultural norms, gender roles. As such, instrumental activities tend to include a broad range of activities.
  Caregivers are asked to rate the degree to which their family member or loved one can perform a variety of tasks. The assessed activities provide a total score from 0-78. Participants with a lower score indicates greater severity.
Time Frame: Baseline to end of treatment period (12 weeks)
Population: Participants with ADCS-ADL scores at Baseline and 12 weeks (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 7.5mg Buntanetap/Posiphen | 15mg Buntanetap/Posiphen | 30mg Buntanetap/Posiphen
Number analyzed (Participants) | 78 | 80 | 74 | 76
units on a scale | 2.03 (0.811) | -0.14 (0.806) | 1.71 (0.831) | 0.15 (0.822)

4. Other Pre Specified Outcome: Change From Baseline to Week 12 in Plasma Biomarkers
Description: Plasma biomarkers measured:
  Glial fibrillary acidic protein (GFAP), Neurofilament light (NFL), TAR DNA-binding protein 43 (TDP43)
Time Frame: Baseline to the end of treatment period (12 weeks)
Population: Participants with analyzable plasma biomarker samples at Baseline and 12 weeks (intent-to-treat population). Plasma biomarkers were an exploratory endpoint; this analysis only included participants from the 30mg buntanetap/posiphen and placebo groups.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo | 30mg Buntanetap/Posiphen
Number analyzed (Participants) | 71 | 70
pg/ml
  GFAP | 5.5 (74.32) | 2.1 (69.44)
  NFL | 0.4 (6.88) | -2.5 (14.05)
  TDP43: number analyzed (Participants) | 61 | 65
  TDP43 | -467.5 (1474) | -985.1 (4950)

5. Post Hoc Outcome: Change From Baseline to Week 12 in ADAS-Cog11 for Biomarker Positive Participants With Baseline MMSE Scores 21-24
Description: Change in the ADAS-Cog11 score from Baseline to the End of Trial. Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog 11) measures cognitive functions and non-cognitive functions such as mood and behavior. It was designed to measure the cognitive and behavioral domains known to be affected in Alzheimer disease, including memory, language, orientation, construction, and planning of simple designs, and completed simple goal-oriented behaviors.
  Specifically, the ADAS-Cog comprises ratings from 11 components: word recall, word recognition, constructional praxis, orientation, naming objects and fingers, commands, ideational praxis, remembering test instructions, spoken language, word finding, and comprehension.
  Total scores range from 0-70, with higher scores indicating greater cognitive impairment.
Time Frame: Baseline to the end of treatment period (12 weeks)
Population: AD biomarker positive participants (pTau217/t-Tau Ratio ≥4.2%) with Baseline MMSE Scores 21-24 and with ADAS-Cog11 scores at Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 7.5mg Buntanetap/Posiphen | 15mg Buntanetap/Posiphen | 30mg Buntanetap/Posiphen
Number analyzed (Participants) | 18 | 20 | 22 | 22
units on a scale | -0.26 (0.911) | -2.19 (0.865) | -2.79 (0.815) | -3.32 (0.820)

ADVERSE EVENTS:
Time Frame: From consent to end of trial (up to 5 months)
Description: A total of 5 participants were mistakenly randomized in the interactive response technology (IRT) system but did not meet inclusion/exclusion criteria at the time of initial treatment. Therefore, these participants did not receive study drug or placebo and were withdrawn from the study. This is the difference between enrollment/participant flow and the number of participants assessed for adverse events.
Arm/Group | Placebo | 7.5mg Buntanetap/Posiphen | 15mg Buntanetap/Posiphen | 30mg Buntanetap/Posiphen
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/86 | 0/85 | 0/87
Serious Adverse Events (participants affected / at risk) | 3/88 | 0/86 | 0/85 | 3/87
Other Adverse Events (participants affected / at risk) | 1/88 | 5/86 | 1/85 | 1/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | 7.5mg Buntanetap/Posiphen (N=86) | 15mg Buntanetap/Posiphen (N=85) | 30mg Buntanetap/Posiphen (N=87)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=88) | 7.5mg Buntanetap/Posiphen (N=86) | 15mg Buntanetap/Posiphen (N=85) | 30mg Buntanetap/Posiphen (N=87)
Dizziness (Nervous system disorders) | 1 (1) | 5 (6) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Annovis Bio's agreements with its investigators may vary. However, Annovis Bio does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data for a clinical trial or for 12 months.

DOCUMENTS (2):
  • Study Protocol (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT05686044/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT05686044/SAP_001.pdf